CLINICAL TRIAL: NCT01197066
Title: A Phase Ⅲ Multicenter, Open-label, Follow-up Study, to Assess the Safety and Efficacy of Certolizumab Pegol as Additional Medication to Methotrexate, in Patients With Active Rheumatoid Arthritis Who Participated in Study 101-KOA-0801i
Brief Title: Open-label, Extension Study of CDP870 in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101-KOA-0802i
Record Dates: First submitted 2010-03-17; First posted 2010-09-09 (Estimated); Last update posted 2022-06-10 (Actual); Status verified 2017-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Certolizumab Pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Certolizumab Pegol (Other): Single Arm
  Interventions: Drug: Certolizumab Pegol

INTERVENTIONS:
Drug: Certolizumab Pegol — Certolizumab Pegol 200mg
  Other Names: CDP870; CIMZIA; Perstymab

SUMMARY:
This is a phase Ⅲ multicenter, open-label, follow-up study, to assess the safety and efficacy of certolizumab pegol (CZP) as additional medication to methotrexate (MTX), in patients with active rheumatoid arthritis (RA) who participated in Study (Protocol) # 101-KOA-0801i.

ELIGIBILITY:
Inclusion Criteria:

* Failed to achieve an ACR20 response at Week 12 in the Study 101-KOA-0801i or completed the entire Study 101-KOA-0801i through Week 24
* Have a clear chest X-ray at the Entry visit
* Negative urine pregnancy test at the Entry
* Continue treatment on methotrexate

Exclusion Criteria:

* Any other inflammatory arthritis (e.g., psoriatic arthritis, ankylosing spondylitis or reactive arthritis)
* Secondary, non-inflammatory type of arthritis (eg, osteoarthritis, fibromyalgia)
* At study entry taking any of the prohibited medications as detailed in the Study (Protocol) # 101-KOA-0801i
* NYHA (New York Heart Association) Class III or IV congestive heart failure
* Current or history of tuberculosis
* History of chronic infection, recent serious or life-threatening infection or any current sign or symptom that may indicate an infection (e.g., fever, cough)
* History of a lymphoproliferative disorder including lymphoma or signs and symptoms suggesting lymphoproliferative disease
* High risk of infection
* Female breast feeding, pregnant or plan to become pregnant during the trial or for 12 weeks following the last dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2010-03 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
To assess the safety of CZP for a long term period as additional medication to MTX, in patients with active RA, as measured by adverse events frequency, severity and nature; PE and vitals; and laboratory values, blood parameters and urine parameters. | Up to 7 years
  Treatment will continue until the drug is commercially available in the country.

SECONDARY OUTCOMES:
To assess the clinical response rate measured by ACR20, ACR50 and ACR70 responder rate. | Up to 7 years
  Treatment will continue until the drug is commercially available in the country.
Improvement in patient's Health-Related Quality of Life (HRQOL) as measured by the 36-item Short Form Health Survey (SF-36) | Up to 7 years
  Treatment will continue until the drug is commercially available in the country.
To assess the achievement of clinical remission measured by DAS28. | Up to 7 years
  Treatment will continue until the drug is commercially available in the country.
The improvement in physical function as measured by the Health Assessment Questionnaire Disability Index (HAQ-DI). | Up to 7 years
  Treatment will continue until the drug is commercially available in the country.

CONTACTS AND LOCATIONS:
Overall Officials: YoungMo Kang, MD, PhD, Principal Investigator — Kyungpook National University Hospital